CLINICAL TRIAL: NCT00535340
Title: An Eight-Week, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Fixed Dose of SR58611A 350 mg Twice a Day in Elderly Patients With Generalized Anxiety Disorder With an Optional Twenty-Four Week Extension
Brief Title: An Eight-Week Study to Evaluate the Efficacy and Safety of SR58611A in Elderly Patients With Generalized Anxiety Disorder
Acronym: GEMINI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: reprioritization of indications
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5895; EudraCT 2006-004147-33
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Anti-Anxiety Agents
MeSH Terms: conditions — Anxiety Disorders | interventions — Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR58611A

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of SR58611A 350 mg twice a day compared to placebo in elderly patients with Generalized Anxiety Disorder (GAD), as assessed by the 14-item Hamilton Anxiety rating Scale (HAM-A).

Secondary objectives are to evaluate the tolerability and safety of SR58611A in elderly patients with GAD, to evaluate the efficacy of SR58611A compared to placebo on disablility and quality of life in elderly patients with GAD and to evaluate the tolerability and safety of 24 weeks of additional treatment with SR58611A in elderly patients with GAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Generalized Anxiety Disorder (GAD) as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria and supported by the Mini International Neuropsychiatric Interview (MINI) plus Generalized Anxiety Disorder module

Exclusion Criteria:

* Minimum total score of less than 22 on the 14-item HAM-A scale
* Total score of 18 or higher on the Montgomery-Asberg Depression Rating Scale (MADRS)
* Mini-Mental State Examination (MMSE) score of 22 or less

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to visit 7 (Day 56) in the 14-item Hamilton Anxiety Rating Scale (HAM-A) total score

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) Severity of Illness Score
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com